CLINICAL TRIAL: NCT00601302
Title: A Single Dose, Two-Period, Two-Treatment, 2-Way Crossover Bioequivalency Study of 10 mg Amlodipine Besylate Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Amlodipine Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMLO-02
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Hypertension; Chronic Stable Angina; Vasospastic Angina
MeSH Terms: conditions — Hypertension; Angina, Stable; Angina Pectoris, Variant | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Amlodipine

SUMMARY:
The objective of this study was the bioequivalence of a Roxane Laboratories' Amlodipine Besylate tablets, 10 mg, to Norvasc® Tablets, 10 mg (Pfizer) under fed conditions using a single-dose, randomized, 2-treatment, 2-period, 2-sequence crossover design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to Amlodipine Besylate or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-04; Primary Completion 2004-04 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Twenty-one day washout

CONTACTS AND LOCATIONS:
Overall Officials: Walter Parham, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States